CLINICAL TRIAL: NCT04371835
Title: COVID-19 in People Living With HIV: Evaluation of Risk Factors and Outcomes in Resource-limited Settings. A Pooled Substudy of ADVANCE, D²EFT, DolPHIN2 and NAMSAL
Brief Title: COHIVE: Coronavirus (COVID-19) Outcomes in HIV Evaluation in Resource Limited Settings
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: University of Witwatersrand, South Africa (Other); University of Liverpool (Other); Université Montpellier (Other); UNITAID (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-04-COHIVE
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: HIV-infection/Aids; Coronavirus Infection
Keywords: Covid-19; SARS-CoV-2; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COHIVE is an observational cohort nested in four antiretroviral therapy research studies (ADVANCE - NCT03122262; D²EFT - NCT03017872; DolPHIN2 - NCT03249181 and NAMSAL-ANRS12313 - NCT02777229). COHIVE will include participants who are possible COVID-19 cases with symptoms or confirmed COVID-19 cases, and participants who agree to have a serology testing for SARS-CoV-2 regardless of COVID-19 history.

DETAILED DESCRIPTION:
COHIVE is an observational cohort study nested within four parent open label randomised clinical trials of first- and second-line antiretroviral therapies (ADVANCE - NCT03122262; D²EFT - NCT03017872; DolPHIN2 - NCT03249181 and NAMSAL-ANRS12313 - NCT02777229). COHIVE objective is to study the occurrence and outcomes of COVID-19 in people living with HIV across a variety of clinical settings. Taken together, these pivotal trials provide an established population and encompass a range of HIV therapies, HIV populations, and geographic regions to capture the full spectrum of these global public health emergency as it pertains to people living with HIV.

The sample will include participants who are possible symptomatic or confirmed COVID-19 cases, and participants who agree to enrol in the SARS-CoV-2 seroprevalence cohort (regardless of SARS-CoV-2 infection). Approximately 2,500 participants are enrolled in these 4 studies.

Enrolment into COHIVE substudy is voluntary and optional for participants in ADVANCE, D²EFT, DolPHIN2 and NAMSAL studies. Parameters relevant to COHIVE substudy including demographics, arm of randomised ART, medical and HIV history, immunological and virological results, adverse events at required time points will be collected as part of parent studies. Substudy specific assessments performed at baseline include optional sample collection for SARS-CoV-2 RT-PCR and serology; for the possible symptomatic or confirmed COVID-19 cases, the management of the patients, diagnostic test results, and outcomes, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Either: i) Meet local testing criteria for COVID-19, or present with symptoms that in the opinion of the investigator are consistent with COVID-19 and do not have an alternative explanation, or have tested elsewhere and found positive for COVID-19; OR ii) Agree for serology testing for SARS-CoV2, regardless of history of COVID-19.
* Have signed the informed consent of one of the parent study.
* Give informed consent to the COHIVE substudy.

Exclusion Criteria:

* Refuse to participate in the COHIVE substudy.
* Any condition which would place the participant at risk if they participated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The substudy will be proposed to all the sites participating in ADVANCE, D²EFT, DolPHIN2 and NAMSAL studies. This substudy will enrol eligible patients with i) confirmed or suspected infection with SARS-CoV-2 and ii) any participants of the 4 parent studies who accept to enrol in the seroprevalence cohort during a scheduled parent study protocol visit following control of the epidemic in country.
Sampling Method: Non-Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical features of symptomatic COVID-19 in people living with HIV (PLWH) | At baseline
  To characterise the clinical features of symptomatic COVID-19 in PLWH (cardio-respiratory and other clinical signs or symptoms), described overall and by HIV and comorbid disease factors including pregnancy status.
Clinical outcomes of symptomatic COVID-19 in PLWH | At Day 28
  To characterise the clinical outcomes of symptomatic COVID-19 in PLWH, assessing the outcomes of patients including the percentage of patients who are fully recovered, required hospitalisation, developed severe illness (ICU admission or equivalent) or died.
Clinical outcomes of symptomatic COVID-19 in PLWH | At Month 3
  To characterise the clinical outcomes of symptomatic COVID-19 in PLWH, assessing the outcomes of patients including the percentage of patients who are fully recovered, required hospitalisation, developed severe illness (ICU admission or equivalent) or died.

SECONDARY OUTCOMES:
Seroprevalence of COVID-19 in all parent study participants | Through study completion, an average of one year
  To determine seroprevalence of COVID-19 in all parent study participants regardless of COVID-19 history.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Calmy, MD, PhD, Principal Investigator — University Hospital, Geneva; Eric Delaporte, MD, PhD, Principal Investigator — IRD, Inserm, University of Montpellier; Saye Khoo, MD, PhD, Principal Investigator — University of Liverpool; Emmanuelle Papot, MD, Principal Investigator — Kirby Institute; Mark Polizzotto, MD, PhD, Study Chair — Kirby Institute; Francois WD Venter, MD, Principal Investigator — Wits Reproductive Health and HIV Institute; Joana Woods, MD, Principal Investigator — Wits Reproductive Health and HIV Institute
Locations (15):
- Hospital G de Agudos JM Ramos Mejia, Buenos Aires, Buenos Aires F.D., Argentina
- Laboratório de Pesquisa Clinica Em Hiv/Aids - Instituto Nacional de Infectologia - Fiocruz, Rio de Janeiro, Brazil
- Cameroon (3):
  - Central Hospital of Yaoundé, Yaoundé
  - Cité Verte Hospital, Yaoundé
  - Hôpital Militaire de Région N°1, Yaoundé
- CART CRS, VHS Hospital, Chennai, Tamil Nadu, India
- Univerity of Malaya Medical Centre, Kuala Lumpur, Malaysia
- Institute of Human Virology, Nigeria (IHVN), Abuja, Nigeria
- South Africa (4):
  - Desmond Tutu HIV Foundation, Cape Town
  - Perinatal HIV Research Unit (PHRU), Johannesburg
  - Clinical HIV Research Unit (CHRU), Wits Health Consotium (Pty) Ltd, Johannesburg
  - Ezintsha, Parktown
- HIV-NAT (The HIV Netherlands Australia Thailand Research Collaboration), Thai Red Cross AIDS Research Centre, Bangkok, Thailand
- Infectious Diseases Institute, Kampala, Uganda
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided